CLINICAL TRIAL: NCT03454880
Title: Measuring Physical Activity Levels in Critical Care: A Feasibility Study
Brief Title: Measuring Physical Activity Levels in Critical Care
Acronym: ACTIVE
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18IR06
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Critical Care
Keywords: Accelerometry; Wearable electronic devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be a single-centre, prospective observational study to evaluate the use of a wearable accelerometer device to measure physical activity levels of patients within critical care.

DETAILED DESCRIPTION:
The study will be a single-centre, prospective observational study involving patients admitted to critical care.

The study is a feasibility study to evaluate the use of a wearable accelerometer device within critical care.

The study participants will be patients admitted to a single critical care unit. Screening of new admissions will be completed and participants recruited according the the inclusion/exclusion criteria.

Participants will not be expected to do anything different to normal as part of the study except wear an accelerometer device on their thigh for the duration of their critical care admission. This will be applied to the patient by the principle investigator, clinical supervisor or member of the critical care research team, as soon as possible after admission. This will take place on the critical care unit and will not require the patient to be moved. The device will be placed on the participant's right thigh unless this is prohibited by lines, wounds or dressings when it will be placed on the left thigh. The device will be covered in a waterproof dressing so that it will not need to be removed during routine personal care. All devices will be fully charged and calibrated prior to application.

In addition, once the device is fitted, the critical care the nursing staff looking after the participant will fill out a simple record sheet each hour during the day shift to document the participant's activity. The activity observation data collection sheet will be based on one previously used in a United Kingdom research study. This data is routinely collected by physiotherapists on the unit at each therapist-patient contact but is not routinely collected hourly by the nursing staff. Recording observed activity will be performed to further explore the feasibility of the data collected from the wearable device.

A priori criteria for feasibility success are recommended by the Consolidated Standards of Reporting Trials (CONSORT) statement extension for feasibility trials and as such a wear time of 10 hours per day and at least 3 days of data will be considered as the criteria for feasibility success.

Due to the nature of this study, the wearable device needs to be fitted within the first 24 hours following admission to critical care. This allows the feasibility of using the device to be evaluated at all stages of a patient's admission within critical care. It is likely that the patients will have undergone intubation and initiation of mechanical ventilation during this time. These patients will be sedated as part of their medical management and as such will not be able to provide consent prior to inclusion. It may not be appropriate to approach the relatives before the first measurement is taken so consent will be waived until discussed with an appropriate consultee. A consultee will be approached as soon as is appropriate, which will generally be within 48 hours after admission. A consultee will be identified after discussion with the participant's family and friends and will be approached by either the principal investigator or a member of the Critical Care research team. They will be able to advise on the presumed thoughts and wishes of the participant. Consultees will be provided with an information sheet and after an appropriate time will be asked to sign a consultee declaration form. If the consultee does not wish for the patient to be included in the study, any data previously collected will be destroyed.

Once the participant has regained capacity and is able to provide their consent they will be provided with a patient information sheet by the principal investigator or member of the critical care research team. The participant will be allowed adequate time (at least 24 hours) for consideration prior to signing a participant re-consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. 'At risk' of physical morbidity as determined by National Institute for Health and Care Excellence (NICE) Clinical Guideline 83
3. Advice from consultee for participation and patient re-consent if appropriate for continuing participation

Exclusion Criteria:

1. Age <18
2. Expected to die during admission
3. Failure to obtain consent or advice,
4. Pre-existing neuromuscular disease
5. Unable to wear accelerometer device
6. Open abdomen
7. Active neurological event requiring intervention (e.g. External Ventricular Drain, Intracranial Pressure bolt)
8. Acute spinal cord injury
9. Lower extremity fractures
10. Bedbound prior to admission

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be patients admitted to University Hospital Wales critical care unit. It is a 33 bedded mixed unit, providing tertiary care for patients from across South and West Wales. Nursing care is provided 1:1 for level 3 care and 1:2 for level 2 care. Patients present with a wide range of medical conditions including post-surgery, polytrauma, respiratory failure and neurological injury. The severity of illness will be variable, but patients admitted to critical care will require support for at least one organ. The majority of patients are likely to be sedated and mechanically ventilated on admission to the unit or shortly afterwards. Patients at high risk of developing physical morbidity will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Wear time | Until discharge from critical care, up to 12 weeks maximum.
  Amount of time device worn (hours per day)
Number of days worn | Until discharge from critical care, up to 12 weeks maximum.
  Number of days worn for at least minimum requirement (10 hours per day)
Number of adverse events | Until discharge from critical care, up to 12 weeks maximum.
  Number of adverse events occuring during device wear
Percentage agreement with observation | Until discharge from critical care, up to 12 weeks maximum.
  Percentage of activities observed by nursing staff recorded by device

SECONDARY OUTCOMES:
Time spent performing activity | Until discharge from critical care, up to 12 weeks maximum.
  Amount of time spent performing activity (minutes/hours)
Time spent in chair | Until discharge from critical care, up to 12 weeks maximum.
  Amount of time spent sitting in chair (minutes/hours)
Time spent in bed | Until discharge from critical care, up to 12 weeks maximum.
  Amount of time spent in bed (minutes /hours)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Jones, Principal Investigator — Student
Locations (1):
- Univeristy Hospital Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connolly BA, Mortimore JL, Douiri A, Rose JW, Hart N, Berney SC. Low Levels of Physical Activity During Critical Illness and Weaning: The Evidence-Reality Gap. J Intensive Care Med. 2019 Oct;34(10):818-827. doi: 10.1177/0885066617716377. Epub 2017 Jul 4. PMID 28675113

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03454880/Prot_SAP_000.pdf
  • Informed Consent Form: Consultee declaration form (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03454880/ICF_001.pdf
  • Informed Consent Form: Participant re-consent form 1 (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03454880/ICF_002.pdf
  • Informed Consent Form: Participant re-consent form 2 (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03454880/ICF_003.pdf